CLINICAL TRIAL: NCT06571994
Title: Examining the Effect of Minimal Plastics Exposure on Plastic-Associated Chemicals (PAC) Excretion and Biomarkers in Adults With Cardiometabolic Risk Factors
Brief Title: The Plastic Exposure Reduction Transforms Health Trial
Acronym: PERTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Western Australia (Other)
Collaborators: The Minderoo Foundation (Unknown)
Responsible Party: Principal Investigator, Michaela Lucas, Professor, The University of Western Australia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021_ET001118
Record Dates: First submitted 2024-07-31; First posted 2024-08-26 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Endocrine Disruptors; Inflammation; Cardiometabolic Risk Factors
Keywords: Plastic; Microplastic; Nanoplastic; Plastic associated chemicals; Bisphenols; Phthalates; Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Masking Description: The statisticians and laboratory personnel involved in analysis of the biological samples will be blinded to participant status
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Plastic Intervention Group (Experimental): 30 participants randomly assigned to the intervention group will consume low PAC food, employ low risk PAC food preparation practices, and use low PAC personal care and cleaning products.
  Interventions: Behavioral: Low Plastic Intervention
- Control Group (No Intervention): 30 participants randomly assigned to the control group will not receive the intervention nor expected to change behaviour.

INTERVENTIONS:
Behavioral: Low Plastic Intervention — Participants will be provided with food that contain no or low plastic and PAC. This is defined as minimally processed (according to NOVA Classification) fresh produce where the supply chain is either known to be free, or likely to be free of plastic contamination. Foods that are canned, pickled, use plastic storage containers will be either avoided or substituted where possible with glass. Participants will also follow guidance concerning the preparation of their food. Plastic utensils used in the preparation of food will be substituted for non-plastic. Commonly used personal care products, e.g., shampoo and soaps, and cleaning products will be replaced with no/low PAC alternatives. Participants will be supplied with a comprehensive schedule, and instructions for the 4-week intervention.
  Arms: Low Plastic Intervention Group

SUMMARY:
The goal of this randomized controlled trial is to learn if an intervention of reducing plastic exposure through diet, personal care and cleaning products can improve health outcomes in adult participants with cardiometabolic risk factors. The main questions it aims to answer are:

* Will the low plastic exposure intervention reduce urinary excretion of bisphenols?
* Will the low plastic exposure intervention reduce urinary excretion of phthalate metabolites?
* Can reducing plastic exposure improve cardiometabolic biomarkers?

Researchers will compare this 4-week low plastic intervention with a control/no intervention group.

Participants in the intervention group will:

* be provided with food that have no/low plastic and plastic-associated chemicals
* be provided with personal care and cleaning produces that have no/low plastic and plastic-associated chemicals
* replace cooking and food preparation equipment with no/low plastic alternatives

Participants in the control group will not receive the intervention and are not expected to change their behaviour.

All participants will provide biological samples (urine, stool, nasal lavage and blood) at several timepoints during the study and attend 4 clinic visits: screening and before, during and after the intervention. Participants will also complete the sociodemographic questionnaire, a physical activity assessment using the International Physical Activity Questionnaire (IPAQ - Short Form), the 24-hr personal care product recall questionnaire, the plastic-associated chemicals questionnaire and be interviewed by a member of the research team to complete a 24-hour diet recall (24DR-PE) of food consumed, and how it was stored prepared, and consumed. The 24DR-PE will facilitate assessments of deviations from the protocol, and enable the assessment of energy, macro and micronutrient intake.

DETAILED DESCRIPTION:
Many plastic products contain endocrine disrupting chemicals, such as bisphenols and phthalates (referred to as plastic-associated chemicals or PAC), which leach out from everyday use and enter the human body. Food contaminated from packaging or with plastic particles, personal care and cleaning products may be sources of PAC which can be inhaled or absorbed through the skin. The fundamental premise underpinning the research is that exposure to PAC, combined with genetic and lifestyle factors, creates chronic and systemic inflammation that underpins cardiometabolic conditions.

This randomized controlled trial aims to demonstrate whether decreasing exposure to plastic and PAC will reduce urinary excretion of PAC and improve cardiometabolic biomarkers in people with cardiometabolic risk factors.

Participants that have consented and passed health screening (N=60) will be randomized to one of two parallel groups, to receive a 4-week low plastic intervention in their homes with the support of registered dietitians.

* Group 1 (N=30): low plastic intervention group
* Group 2 (N=30): control/no intervention group

All participants will attend four in-person clinic appointments, one during screening, and three during the intervention (Visit 1: day 0, baseline; Visit 2: day 16, midpoint; and Visit 3: day 29, post intervention), of up to two hours duration each. In addition, participants will have a video/phone appointment between screening and Visit 1.

The day before and after the video/phone appointment, participants will be asked to collect urine, stool and nasal washing samples and send them back the day after their video/phone appointment. At the end of the video/phone appointment, eligible and willing participants will be invited to continue to the intervention study and randomized into either the intervention or control group. At the video/phone appointment, participants from Group 1 will order their food and personal care products. The researchers will send the order to a local meal service delivery who will order, pay for, package, and deliver the approved food to the participants' homes in insulated boxes. Delivery of approved products to participants' homes will take place the day before the intervention begins, and at other pre-determined timepoints throughout the study, as required. Samples of food products will be frozen for retrospective testing for PAC, if exposure testing indicates contamination from an unexpected source. Participants from Group 1 will use only non-plastic cooking utensils provided by the researchers and follow guidance concerning the preparation of their food. Participants from Group 1 will use only personal care and cleaning products supplied by the research team. Personal care products include, but are not limited to shampoo, conditioners, face moisturizers, cleansers, serums, make-up and sunscreens, deodorant, tampons and applicators. Participants will be supplied with a comprehensive schedule, and instructions for the 4-week intervention.

All participants will be asked to collect urine, stool, and nasal washing samples on days -1, 8, 15, 22 and 28 of the intervention period, and return them at the clinic visits. During the clinic visits, participants will have fasting blood sample taken, complete the sociodemographic questionnaire, a physical activity assessment using the International Physical Activity Questionnaire (IPAQ - Short Form), the 24-hr personal care product recall questionnaire, the plastic-associated chemicals questionnaire and be interviewed by a member of the research team to complete a 24-hour diet recall - plastic exposure (24DR-PE) of food consumed, and how it was stored prepared, and consumed. The 24DR-PE will facilitate assessments of deviations from the protocol, and enable the assessment of energy, macro and micronutrient intake.

For intervention adherence the following assessment tools will be employed:

24-hour dietary recall - plastic exposure interview (24DR-PE): This assessment is a researcher-administered, computer-assisted, 24-hour dietary recall interview. The method assesses dietary intake on the preceding 24-hour period. The method is adapted to gather additional information concerning the packaging, storage, and preparation of food by the participants. Trained dietitians will carry out the interviews during the clinic visits. The interviews will vary in length between 15 and 60 minutes depending on the stage of the study, and the complexity of each participants' diet. They will be carried out once during screening and three times during the 4-week intervention.

24-hour personal care product recall (24HR-PPR): This is a self-administered questionnaire for the 24-hour recall of personal care products use. This assessment will be conducted once during screening and three times during the 4-week intervention. The questionnaire consists of 15 questions and will take between 2 and 5 minutes to complete.

Post-trial survey: This survey will be conducted to identify any difficulties experienced by the participants that might have affected their adherence to the intervention and procedures.

Tolerability and feasibility qualitative interview: To evaluate the tolerability and feasibility of the trial intervention, participants will be invited to participate in a phone interview within two weeks of completing the intervention. A trained interviewer will conduct the interviews using a structured guide that includes both closed and open-ended questions. Each interview is expected to last 20-40 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Biological males or, non-pregnant, non-lactating biological females aged 18 to 60 years.

   a) For female participants at least one of the following must apply: i) Not of childbearing potential - surgical sterile or postmenopausal (no menses last 12 months and follicle-stimulating hormone (FSH) greater than 40 mIU/mL); ii) Childbearing potential and agrees to practice true abstinence, is in a same-sex relationship or agrees to use effective contraception during the study (either hormonal contraception, intrauterine devices or condom) or has a vasectomised male partner.
2. Body mass index ≥30 kg/m2. If outside this range, eligible at investigator's discretion.
3. Waist circumference ≥102cm in men and ≥88cm in women. If outside this range, eligible at investigator's discretion.
4. Certain medications may be excluded based on investigators discretion.
5. Lives in the Perth Metropolitan Area.
6. Willing to change all they eat, not eat out and not wear makeup for 4 weeks if selected for intervention.
7. Ability to give written informed consent.
8. Proof of immunisation against COVID-19 (SARS-CoV-2), according to WA Health guidelines at time of recruitment.

Exclusion Criteria:

1. Any abnormalities in electrocardiogram (ECG) readings, or as per the Investigator's discretion.
2. History of drug or alcohol abuse in the past 24 months. Alcohol abuse defined as greater than 21 units/week for males, greater than 14 units/week for females.
3. Current regular smoker or e-cigarette use. Social smokers (less than 3 nicotine/tobacco products in the last 3 months) can be included if abstaining for the duration of the study.
4. Currently pregnant or planning pregnancy during the course of the study as assessed by pregnancy testing carried out during screening.
5. Currently on, or within 3 months of discontinuing, glucagon-like peptide-1 agonists or related compounds. If inside this range, eligible at Investigator's discretion.
6. Living in a home that has been renovated in the past 4-weeks.
7. Have known severe food allergies or anaphylaxis to common food allergens. As per the Investigator's discretion.
8. Not suitable for the study for any other reason, as determined by the investigator.
9. Acute infection, surgery, vaccination, or other inflammatory process in the previous 2 weeks. Minor procedures are exempt at investigator's discretion.
10. Evidence of moderate or greater renal impairment at screening, as indicated by an estimated creatinine clearance of less than 60 mL/min using the Cockcroft-Gault equation.
11. Clinically significant abnormal laboratory tests or examination findings, as determined by the investigator, not otherwise mentioned.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-07-04 (Actual)

PRIMARY OUTCOMES:
Change in bisphenols (composite of bisphenol A, BPA; and bisphenol S, BPS) | Baseline and 4 weeks for both groups
  Assessed by measuring urinary concentrations (ng/mL) of BPA and BPS and comparing mean percent change

SECONDARY OUTCOMES:
Change in bisphenol A (BPA) | Baseline, and 1, 2, 3 and 4 weeks for both groups
  Assessed by measuring urinary concentrations BPA (ng/mL) and compare mean percent change
Change in bisphenol S (BPS) | Baseline, and 1, 2, 3 and 4 weeks for both groups
  Assessed by measuring urinary concentrations of BPS (ng/mL) and compare mean percent change
Change in diethyl phthalate (DEP) | Baseline, and 1, 2, 3 and 4 weeks for both groups
  Assessed by measuring urinary concentrations (ng/mL) of DEP metabolite, mono-ethyl phthalate (MEP), and compare mean percent change
Change in di-n-butyl-phthalate (DnBP) | Baseline, and 1, 2, 3 and 4 weeks for both groups
  Assessed by measuring urinary concentrations (ng/mL) of DnBP metabolites, mono-n-butyl-phthalate (MnBP) and mono-(3-carboxypropyl) phthalate (MCPP), and compare mean percent change
Change in di-iso-butyl phthalate (DiBP) | Baseline, and 1, 2, 3 and 4 weeks for both groups
  Assessed by measuring urinary concentrations (ng/mL) of DiBP metabolite, mono-iso-butyl phthalate (MiBP), and compare mean percent change
Change in benzyl butyl phthalate (BBP) | Baseline, and 1, 2, 3 and 4 weeks for both groups
  Assessed by measuring urinary concentrations (ng/mL) of BBP metabolite, mono-benzyl phthalate (MBzP), and compare mean percent change
Change in di-(2-ethylhexyl) phthalate (DEHP) | Baseline, and 1, 2, 3 and 4 weeks for both groups
  Assessed by measuring urinary concentrations (ng/mL) of the composite of DEHP metabolites (mono-2-ethylhexyl phthalate, MEHP; mono-(2-ethyl-5-oxohexyl) phthalate, MEOHP; mono-(2-ethyl-5-hydroxyhexyl) phthalate, MEHHP; and mono-(2-ethyl-5-carboxypentyl) phthalate, MECPP) and compare mean percent change

OTHER OUTCOMES:
Changes in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) | Baseline, and 2 and 4 weeks for both groups
  Assessed by measuring glucose (mmol/L) x insulin (mU/L / 22.5 in fasting blood samples
Changes in fasting serum triglycerides | Baseline, and 2 and 4 weeks for both groups
  Assessed by measuring triglycerides (mmol/L) in fasting blood samples
Changes in high sensitivity C-reactive protein (hsCRP) | Baseline, and 2 and 4 weeks for both groups
  Assessed by measuring hsCRP (mg/L) in fasting blood samples
Changes in cholesterol | Baseline, and 2 and 4 weeks for both groups
  Assessed by measuring low-density lipoprotein cholesterol (LDL-C; mmol/L), high-density lipoprotein cholesterol (HDL-C; mmol/L) and remnant cholesterol (mmol/L) in fasting blood samples
Changes in liver function | Baseline, and 2 and 4 weeks for both groups
  Assessed by measuring fasted alanine transaminase (ALT) and aspartate transaminase (AST) in blood samples
Changes in renal function | Baseline, and 2 and 4 weeks for both groups
  Assessed by measuring estimated glomerular filtration rate (mL/min/1.73 m2) using age, sex and plasma/serum creatinine
Changes in adiponectin/leptin ratio | Baseline, and 2 and 4 weeks for both groups
  Assessed by measuring adiponectin and leptin levels (pg/mL) in fasting blood samples
Changes in body composition | Baseline, and 2 and 4 weeks for both groups
  Assessed by measuring mass, fat free mass, visceral adipose tissue, and skeletal muscle mass
Changes in waist circumference | Baseline, and 2 and 4 weeks for both groups
  Assessed by using a non-stretchable tape measure to obtain waist circumference
Changes in blood pressure | Baseline, and 2 and 4 weeks for both groups
  Assessed by measuring systolic/diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Lucas, Principal Investigator — The University of Western Australia
Locations (1):
- Harry Perkins Institute of Medical Research, Nedlands, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No
At this stage of the study the investigators do not plan to share IPD but this decision may be reviewed in the future.

REFERENCES:
- [Derived] Lucas A, Harray A, Duong L, Herrmann S, Vlaskovsky P, Trevenen M, Chan D, Papendorf H, Smith T, Flint L, Liu A, Gaudieri S, Wang X, Mueller JF, Thomas KV, Murray K, Symeonides C, Dunlop S, Watts G, Lucas M. Randomised controlled trial of a low plastic diet and lifestyle intervention for adults with cardiometabolic risk factors: the Plastic Exposure Reduction Transforms Health (PERTH) trial - a protocol. BMJ Open. 2025 Aug 25;15(8):e099330. doi: 10.1136/bmjopen-2025-099330. PMID 40854835